CLINICAL TRIAL: NCT01529359
Title: Effect of Lactibiane Tolerance on Symptoms Severity of Irritable Bowel Syndrome
Brief Title: Irritable Bowel Syndrome and Lactibiane Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Organization: Larena SAS (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PiLeJe-LactiTol-0210
Record Dates: First submitted 2011-10-10; First posted 2012-02-08 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Probiotics Excipients
  Interventions: Dietary Supplement: Placebo
- Lactibiane Tolerance (Experimental): Probiotics combination
  Interventions: Dietary Supplement: Lactibiane Tolerance

INTERVENTIONS:
Dietary Supplement: Lactibiane Tolerance — Probiotics combination 2 gelules per days during 6 weeks
  Other Names: Probiotic
  Arms: Lactibiane Tolerance
Dietary Supplement: Placebo — Placebo 2 gelules per days for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of a probiotic combination (Lactibiane Tolerance) on the severity of symptoms in patients with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the effects of a probiotic combination (Lactibiane Tolerance) on the severity of symptoms in patients with irritable bowel syndrome (IBS).

The secondary purposes are to evaluate the effects of the intervention on:

* quality of life
* severity of fatigue, anxiety and depression
* levels of inflammatory markers in blood and tools

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome according to the Rome II criteria
* 150< Francis Score < 300
* HAD score inferior or egal to 25

Exclusion Criteria:

* History of hypersensitivity to one of the composant of the product
* Use of probiotics or antibiotics last four weeks
* use of prohibited drugs
* bowel preparation for morphological examination last month
* pregnancy or lactation
* immundepressed or co-existing other serious illness or evolutive

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-03-24 (Actual); Primary Completion 2013-02-04 (Actual); Study Completion 2013-02-11 (Actual)

PRIMARY OUTCOMES:
Severity of bowel symptoms according to the Francis Score | After 6 weeks of complementation
  The severity of bowel symptoms is evaluated with a quality of life questionnaire, the Francis Score before and after 6 weeks of complementation in placebo and verum groups.

SECONDARY OUTCOMES:
Quality of life | after 6 weeks of complementation
  Effect of the intervention on transit and abdominal pain
Severity of Anxiety/Depression | after 6 weeks of complementation
  The level of anxiety/depression will be measured with the HAD scale
Impact of the complementation on fatigue | after 6 weeks of complementation
  The level of fatigue will be measured with the score to the fatigue Impact Scale (FIS)
Impact of the intervention on immunological parameters in stools | after 6 weeks of complementation
  The effects of the intervention on immunological parameters in stools will be evaluated via the levels of beta-defensine 2 and sérine protease activities
Impact of the intervention on immunological parameters in blood | after 6 weeks of complementation
  The impact of the intervention on immunological parameters in blood will be measured with levels of endotoxines, ultrasensitive protein C Reactive and cytokines
Severity of bowel symptoms according to the Francis Score | after 2 weeks of wash-out
  The severity of bowel symptoms is evaluated with the Francis Score before 6 weeks of complementation and after 2 weeks of wash-out in placebo and verum groups
Quality of life | after 2 weeks of wash-out
  Effect of the intervention on transit and abdominal pain
severity of the anxiety/depression | after 2 weeks of wash-out
  The level of anxiety/depression will be measured with the HAD scale
Impact of the complementation on fatigue | After 2 weeks of wash out
  The level of fatigue will be measured with the score to the fatigue Impact Scale (FIS)
Impact of the intervention on immunological parameters in stools | after 2 weeks of wash out
  The effects of the intervention on immunological parameters in stools will be avaluated via the levels of beta-defensine 2 and sérine protease activities
Impact of the intervention on immunological parameters in blood | after 2 weeks of wash-out
  The impact of the intervention on immunological parameters in blood will be measured with levels of endotoxines, ultrasensitive protein C Reactive and cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Piche Thierry, MD, Principal Investigator
Locations (1):
- Chu L'Archet 2, Nice, Alpes Maritimes, France